CLINICAL TRIAL: NCT07391072
Title: Bridging the Gap: A Multiple Baseline Design Study on the Effectiveness of a Mobile-based Stress Management Intervention in Adults on Waiting Lists for Mental Healthcare
Brief Title: Effectiveness of a Waitlist App "Stappvoorstap" During Mental Healthcare Waiting Times
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GGZ Centraal (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Sevda Demirel, PhD Candidate, GGZ Centraal
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Stappvoorstap_N24.084; KPO-79 (Other Grant/Funding Number: Zorgondersteuningsfonds)
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Psychological Stress; Coping Ability; Mental Health; Quality of Life; Coping Skills
Keywords: waiting list; mental health; stress management; mobile health; self-management; mHealth; ecological momentary intervention; single-case experimental design; perceived stress
MeSH Terms: conditions — Stress, Psychological; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: 3-week baseline (Experimental): Participants receive 3 weeks of baseline measurements, 4 weeks of Stappvoorstap app intervention, and 3 weeks of follow-up (10 total measurements).
  Interventions: Behavioral: Stappvoorstap: mobile self-management waitlist intervention
- Group 2: 4-week baseline (Experimental): Participants receive 4 weeks of baseline measurements, 4 weeks of Stappvoorstap app intervention, and 3 weeks of follow-up (11 total measurements).
  Interventions: Behavioral: Stappvoorstap: mobile self-management waitlist intervention
- Group 3: 5-week baseline (Experimental): Participants receive 5 weeks of baseline measurements, 4 weeks of Stappvoorstap app intervention, and 3 weeks of follow-up (12 total measurements).
  Interventions: Behavioral: Stappvoorstap: mobile self-management waitlist intervention

INTERVENTIONS:
Behavioral: Stappvoorstap: mobile self-management waitlist intervention — Stappvoorstap is a free mobile self-management application developed in co-creation with mental health waitlist clients. The app measures daily stress levels 2-4 times per day through short questionnaires, creates visual overviews of personal stress patterns on daily and weekly scales, provides real-time coping suggestions, offers mindfulness and relaxation exercises (breathing exercises, meditation, nature sounds, calming music), and includes informational articles and personal experience stories.

SUMMARY:
This study evaluates the effectiveness of Stappvoorstap, a mobile self-management application designed for adults on mental health waiting lists in the Netherlands. The app helps users monitor daily stress levels, recognize personal stress patterns, and provides coping strategies, relaxation exercises, and supportive resources. Using a multiple baseline single-case experimental design, participants use the app for 4 weeks while completing weekly questionnaires measuring perceived stress, coping self-efficacy, and quality of life. The study aims to determine whether the app can reduce stress and improve wellbeing during the waiting period before mental healthcare treatment begins.

DETAILED DESCRIPTION:
Prolonged waiting times for mental healthcare pose significant challenges, with nearly 100,000 people on waiting lists in the Netherlands as of December 2023. During this period, symptoms can worsen, daily functioning may decline, and quality of life decreases. Stappvoorstap was developed in co-creation with waitlist clients and experts-by-experience to address this gap. The app is based on stress-signaling plans used in Dutch mental healthcare and functions as an ecological momentary intervention. It measures perceived stress 2-4 times daily, creates visual overviews of stress patterns, and provides real-time coping suggestions, mindfulness exercises, informational articles, and personal stories from other clients. This study uses a nonconcurrent multiple baseline design with A-B-A design. Participants are randomly assigned to 3, 4, or 5-week baseline phases, followed by 4 weeks of app use, and 3 weeks of follow-up. Weekly assessments include the Perceived Stress Scale (PSS-10), Coping Self-Efficacy Scale (CSES-13), and WHOQOL-BREF. Both group-level and individual case analyses will be conducted using mixed-effects modeling and Tau-(BC) effect size measures.

Participants are recruited from mental health waiting lists across the Netherlands. As this is a mobile app-based intervention, participation is location-independent and takes place remotely.

ELIGIBILITY:
Inclusion Criteria:

* Currently on a waiting list at a mental health organization in the Netherlands.
* Aged 18 years or older
* Owns a smartphone and has the ability to operate it
* Sufficient proficiency in Dutch or English language (at least B1 level)

Exclusion Criteria:

* Currently enrolled in another medical-scientific research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Stress | Weekly measurements for 10-12 weeks (depending on group assignment)
  Measured using the Perceived Stress Scale with 10 items (PSS-10). The PSS-10 is a validated self-report questionnaire assessing how stressful situations were perceived in the past week. Items are rated on a 5-point scale (1=never to 5=very often). Higher scores indicate higher perceived stress. Change from baseline phase to intervention phase, and to follow-up will be assessed.

SECONDARY OUTCOMES:
Change in Coping Self-Efficacy | Weekly measurements for 10-12 weeks (depending on group assignment)
  Measured using the Coping Self-Efficacy Scale with 13 items (CSES-13). The CSES-13 measures confidence in coping behaviors across three subscales: problem-focused coping, emotion-focused coping, and social support coping. Items are rated on a 10-point scale (0=cannot do at all to 10=certainly can do). Higher scores indicate greater coping self-efficacy.
Change in Quality of Life | Weekly measurements for 10-12 weeks (depending on group assignment)
  Measured using selected domains of the World Health Organization Quality of Life Brief version (WHOQOL-BREF): physical health (7 items), psychological health (6 items), and social relationships (3 items), plus 2 items on overall quality of life and general health. Items rated on 5-point Likert scales. Higher scores indicate better quality of life.

OTHER OUTCOMES:
User Experience and Perceived Usefulness | After completion of the 4-week intervention period
  Semi-structured interview assessing participants' experiences with the Stappvoorstap app, including perceived usefulness, usability, barriers and facilitators, and suggestions for improvement. Open-ended questions explore how participants integrated the app into daily life and their overall satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- GGZ Centraal, Almere Stad, Flevoland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Anonymized group-level data may be made available upon reasonable request to the principal investigator, in accordance with institutional and ethical guidelines.

REFERENCES:
- See also: Official website with information about the Stappvoorstap app, and resources for people on mental health waiting lists. — https://stappvoorstap.nl